CLINICAL TRIAL: NCT06604325
Title: Prophylactic Role Of Tranexamic Acid To Reduce Blood Loss During Caesarean Delivery : A Prospective Study.
Brief Title: Prophylactic Tranexamic Acid To Reduce Blood Loss During Caesarean Delivery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aligarh Muslim University (Other)
Responsible Party: Principal Investigator, MUAZZAM HASAN, Associate Professor, Aligarh Muslim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEC-812
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): All women recruited to Group A will receive tranexamic acid 1 gram in 100 ml Normal Saline as intravenous infusion 10 minutes before the skin incision.
  Interventions: Drug: Tranexamic acid injection
- Group B (Placebo Comparator): All women recruited to Group A will receive 100 ml Normal Saline as intravenous infusion 10 minutes before the skin incision, as placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid injection — All women recruited to Group A will receive tranexamic acid 1 gram in 100 ml Normal Saline as intravenous infusion 10 minutes before the skin incision.
  Arms: Group A
Drug: Placebo — All women recruited to Group B will receive 100 ml Normal Saline as intravenous infusion 10 minutes before the skin incision.
  Arms: Group B

SUMMARY:
Postpartum hemorrhage continues to be the leading cause of maternal morbidity and mortality. Globally, it is responsible for 25% of all pregnancy-related deaths. PPH is unpredictable and may occur in the absence of risk factors. Tranexamic acid is an antifibrinolytic proven to reduce blood loss and transfusion requirements for various surgeries. This study aims to explore the effectiveness of tranexamic acid as an adjunct to other uterotonics before the Caesarian Section.

ELIGIBILITY:
Inclusion Criteria:

1. The women undergoing cesarean delivery (both elective and emergency) during the study period.
2. Willing to participate in the study after understanding the concept.

Exclusion Criteria:

1. Critically ill patient.
2. Not willing to give consent to participate in the study
3. Cases diagnosed with a ruptured uterus or undergoing caesarian hysterectomy during operation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women posted for elective or emergency caesarean section.
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood loss | Amount of blood loss from starting from surgical incision till 24 hours post caesarean section.
  The primary aim of the trial is to investigate the effect of tranexamic acid on peri and post- operative blood loss during caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: MUAZZAM HASAN, MD, Principal Investigator — AMU
Locations (1):
- ASJSATDS Medical College, Fatehpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No